CLINICAL TRIAL: NCT07223294
Title: A Randomized, Multicenter, Multiple-dose, Double-blind, Placebo-controlled, Parallel-group Design, Clinical Endpoint Bioequivalence Study to Evaluate the Therapeutic Equivalence and Safety of Fluticasone Furoate and Vilanterol Inhalation Powder 100 mcg/25 mcg (Sandoz) and BREO® ELLIPTA® (Fluticasone Furoate and Vilanterol Inhalation Powder) 100 mcg/25 mcg (GlaxoSmithKline) in Adult Participants With Asthma
Brief Title: Study to Evaluate the Therapeutic Equivalence and Safety of Fluticasone Furoate and Vilanterol Inhalation Powder 100 mcg/25 mcg and BREO ELLIPTA 100 mcg/25 mcg in Participants With Asthma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAN-1138
Record Dates: First submitted 2025-10-15; First posted 2025-10-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Respiratory
MeSH Terms: interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fluticasone furoate and vilanterol inhalation powder (Experimental): Fluticasone furoate and Vilanterol inhalation powder 100 mcg/25 mcg QD for 4 weeks
  Interventions: Combination Product: Fluticasone furoate and vilanterol inhalation powder
- Breo Ellipta (Active Comparator): Fluticasone furoate and Vilanterol inhalation powder 100 mcg/25 mcg QD for 4 weeks
  Interventions: Combination Product: Breo Ellipta
- Placebo (Placebo Comparator): Placebo QD for 4 weeks
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Fluticasone furoate and vilanterol inhalation powder — Fluticasone furoate and vilanterol inhalation powder 100 mcg/25 mcg
  Arms: Fluticasone furoate and vilanterol inhalation powder
Combination Product: Breo Ellipta — Fluticasone furoate and Vilanterol inhalation powder) 100 mcg/25 mcg
  Arms: Breo Ellipta
Combination Product: Placebo — Inhalation powder with lactose
  Arms: Placebo

SUMMARY:
This is a randomized, multi-center, multiple-dose, double-blind, placebo-controlled, Parallel group design, clinical endpoint bioequivalence study in adult participants with asthma.

The study design includes up to a 2-week Screening period, at least a 2-week Run-in period, a 4-week Treatment period, and a safety follow up call one week later.

Visit 1: Screening Visit 2: Run-in period: All eligible participants will enter a 2-week Run-in period in which training will be provided to the participants on the use of inhalers and participant diary.

Visit 3: Day 1: Randomization to one of the 3 treatment groups to receive one inhalation of the study medication quaque die (QD), in the morning, for 28 ± 2 days.

Visit 4: Day 28: EOT

Participants will be contacted one week after their last site visit for Safety follow-up via phone call (end of study). Participants will be instructed to refrain from taking their current inhaled asthma medications from the start of the Run-in period until the end of treatment (EOT) visit. They will be provided with a salbutamol/albuterol inhaler (rescue medication) for use on an as-needed basis during the entire study duration until the EOT visit.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent (as described in the protocol), which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol.
* Participants must be 18 to 75 years old (inclusive) at Screening (signing the ICF).
* Diagnosis of asthma, as defined by the National Asthma Education and Prevention Program, at least 12 weeks prior to Screening.
* Participants who are stable on their chronic asthma treatment regimen for at least 4 weeks prior to Screening.
* Pre-bronchodilator FEV1 of >40% and <85% of predicted value, at Screening.
* Participants with FEV1 reversibility of ≥12% and ≥200 mL within 30 minutes following 360 mcg of albuterol inhalation (via pressurized metered dose inhaler pressurized metered-dose inhaler [pMDI]) or equivalent at Screening.
* This what you mean: Participants who are currently non-smoking and have not used tobacco smoking or smoked marijuana products, within the past year.
* Participants who are able to replace their current regularly scheduled short-acting β2-agonists (SABAs) with a salbutamol/albuterol inhaler for use only on an 'as-needed' basis for the duration of the study.
* Participants must be able to discontinue their asthma medications during the Run-in period, and for the remainder of the study.
* Participants who can demonstrate the correct use of inhaler device (during the Run-in period and at Randomization visit).
* Participants are eligible to participate in this study if they are:
* Of non-childbearing potential
* Of childbearing potential, and if they agree to use a highly effective form of contraception consistently during the study, starting at Screening and until the end of study (EOS). These participants must have a negative pregnancy test at Screening and Randomization visit.
* Participants who produce viable sperm and have a partner of childbearing potential, and if they agree to use an adequate method of contraception consistently during the study, starting at Screening and until the EOS and also refrain from donating sperm during this period. Participants with a partner or partners who is (are) not of childbearing potential are exempt from these requirements.

Exclusion Criteria:

* Participants who have life-threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnia, respiratory arrest or hypoxic seizures, asthma-related syncopal episodes(s), or hospitalizations within one year prior to Screening or during the Run-in period.
* Participants with significant chronic respiratory disease (COPD, interstitial lung disease, etc) other than asthma which in the opinion of the Investigator may interfere with the study evaluation or optimal participation in the study.
* Participants with evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, cardiac dysrhythmia, significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that in the opinion of the Investigator, would put them at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
* Participants with asthma exacerbations (ie, acute or sub-acute worsening in symptoms and lung function from the participant's usual status) within 6 weeks prior to Screening or during the Run-in period.
* Participants with evidence or history of tuberculosis (additionally confirmed with a chest X-ray done within 6 months prior to Screening for countries with high tuberculosis risk).
* Participants with uncontrolled allergic rhinitis within 15 days prior to Screening.
* Viral, bacterial, fungal, or parasitic, acute upper or lower respiratory tract infection (including Coronavirus Disease (COVID-19)), or sinus, or middle ear infection within 4 weeks prior to Screening, during the Run-in period, or at the Randomization visit. Note: Rescreening of participants with acute respiratory conditions during the Screening and Run-in period may be allowed in consultation with Medical Monitor (Section 5.4).
* Participants with a history of hepatitis B, hepatitis C, or human immunodeficiency virus 1 and 2.
* Participants with clinically significant screening laboratory and electrocardiogram (ECG) parameters as per Investigator's assessment.
* Participants receiving systemic, oral, parenteral or depot corticosteroids, or anti-immunoglobulin E (IgE) therapy within 12 weeks prior to Screening spirometry or unable to stop receiving these medications during the study.
* Participants receiving β2-blockers, anti-arrhythmics, anti-depressants, monoamine oxidase inhibitors, cytochrome P450 3 subfamily A member 4 (3A4) inhibitors, or diuretics within 4 weeks prior to the Screening spirometry or unable to stop receiving these medications during the study.
* Participants receiving monoclonal antibodies that may affect the course of asthma within 180 days prior to the Screening spirometry or unable to stop receiving these medications during the study.
* Participants receiving live attenuated vaccines within two days prior to Screening.
* Participants who received an investigational drug within 28 days or 5 half-lives (whichever is longer) prior to Screening.
* Hypersensitivity to any sympathomimetic drug (eg, albuterol, vilanterol) or to any inhaled, intranasal, or systemic corticosteroid therapy, or to milk proteins, or to excipients in the dry powder inhaler.
* Participants with significant alcohol or controlled substance abuse in the past 6 months, per the judgment of the Investigator.
* Participants with any factors (eg, infirmity, disability, or geographic location) that the Investigator feel would likely limit the participants' compliance with the study protocol or scheduled clinic visits.
* Participants who cannot communicate reliably or who are unlikely to co-operate with the requirements of the study, in the opinion of the Investigator.

Participants who are pregnant, breastfeeding, or planning to become pregnant during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1430 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the therapeutic equivalence of test and reference product | Day 1 (0-24Hrs)
  Forced Expiratory Volume in 1 Second (FEV1) Are Under Curve (AUC 0-24) on Day 1
Demonstrate the therapeutic equivalence of test and reference product | Day 28 of treatment
  trough Forced Expiratory Volume in 1 Second (FEV1 on Day 28)
Demonstrate the superiority of test and reference product over placebo | Day 1 (0-24 hours (Hrs)
  Forced Expiratory Volume in 1 Second (FEV1) Are Under Curve (AUC 0-24) on Day 1
Demonstrate the superiority of test and reference product over placebo | Day 28 of treatment
  trough Forced Expiratory Volume in 1 Second (FEV1 on Day 28)

SECONDARY OUTCOMES:
To compare the number and type of Adverse Events of Test, Reference and Placebo | Screening to week 5 (End of study)
  Number of Adverse Events, Serious Adverse Events, Treatment-Emergent Adverse Events (TEAE)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Sandoz Investigational Site, Cullman, Alabama
  - Sandoz Investigational Site, Bradenton, Florida
  - Sandoz Investigational Site, Leesburg, Florida
  - Sandoz Investigational Site, Orlando, Florida
  - Sandoz Investigational Site, St Louis, Missouri
  - Sandoz Investigational Site, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No